CLINICAL TRIAL: NCT06998589
Title: Comparison of the Efficacy and Safety of Delicate Pulsed Light and Q-Switched 1064 nm Nd:YAG Laser in the Treatment of Post-Acne Erythema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, Weihui Zeng, Professor, Second Affiliated Hospital of Xi'an Jiaotong University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025086
Record Dates: First submitted 2025-05-17; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Post-acne Erythema
Keywords: post-acne erythema

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DPL (Experimental): The DPL treatment was randomly applied to one side of the face, with an energy density of 6-8 J/cm². Sessions were performed at intervals of 2-3 weeks, for a total of six treatments.
  Interventions: Other: DPL
- Q-switched 1064 nm Nd:YAG laser (Experimental): The randomly assigned half of the face received large-spot, low-energy 1064 nm laser treatment at an energy density of 0.8-1 J/cm², performed at intervals of 2-3 weeks for a total of six sessions.
  Interventions: Other: DPL

INTERVENTIONS:
Other: DPL — The DPL treatment was randomly applied to one side of the face, with an energy density of 6-8 J/cm². Sessions were performed at intervals of 2-3 weeks, for a total of six treatments..The randomly assigned half of the face received large-spot, low-energy 1064 nm laser treatment at an energy density of 0.8-1 J/cm², performed at intervals of 2-3 weeks for a total of six sessions.

SUMMARY:
Acne vulgaris is a common chronic dermatological condition, affecting approximately 85% of adolescents worldwide and ranking eighth among all chronic diseases. Its exacerbation is often associated with recurrent lesions, inadequate treatment, and poor skincare habits such as squeezing or scratching, which frequently lead to the development of post-acne erythema (PAE). PAE is a vascular lesion located beneath the surface of the skin, characterized by a red appearance due to the clustering of dilated capillaries. Although PAE typically improves within 2 to 6 months, it may persist longer in some cases and even result in post-inflammatory hyperpigmentation. This is particularly prevalent in individuals with darker skin tones, where the incidence of PAE and hyperpigmentation ranges from approximately 45.5% to 87.2%. Facial acne not only affects physical appearance but also significantly impairs social interactions and can lead to psychological distress, including low self-esteem and depression.

Low-energy, large-spot 1064 nm Nd:YAG laser, which belongs to the near-infrared spectrum, has deeper skin penetration and can effectively target deeper dermal tissues. In the treatment of PAE, the laser energy is absorbed by dilated microvasculature in the skin, promoting vasoconstriction and reducing localized redness and swelling. The low energy setting minimizes thermal damage while stimulating collagen production, thereby enhancing skin repair and improving the appearance of erythema.

Delicate Pulsed Light (DPL) operates by emitting pulses of light at specific wavelengths that selectively target skin chromophores. In treating PAE, DPL precisely controls the wavelength and pulse intensity to target dilated blood vessels, thereby alleviating redness and inflammation. Additionally, DPL stimulates the skin's natural repair mechanisms and promotes collagen synthesis, accelerating the resolution of erythema and enhancing overall skin texture. Compared with conventional Intense Pulsed Light (IPL), DPL offers more accurate light modulation, fewer side effects, and better adaptability to various skin types and conditions.

In this study, we conducted a split-face randomized controlled trial to compare the clinical efficacy and safety of low-energy large-spot 1064 nm Nd:YAG laser and DPL in treating acne and PAE. We aimed to explore whether there are significant differences between these two modalities in terms of clinical outcomes for post-acne erythema.

DETAILED DESCRIPTION:
Acne vulgaris is a highly prevalent chronic inflammatory skin disease, affecting approximately 85% of adolescents globally, and ranking eighth among all chronic conditions in terms of global disease burden. Although traditionally perceived as a benign and self-limiting disorder, its impact on quality of life, especially when accompanied by persistent post-lesional sequelae such as post-acne erythema (PAE), is increasingly recognized. The aggravation of acne is often multifactorial, closely linked to recurrent inflammatory episodes, inadequate therapeutic interventions, and improper skincare behaviors such as manual squeezing or scratching of lesions. These factors not only exacerbate active lesions but also contribute significantly to the development and persistence of PAE.

PAE is a vascular response resulting from the dilation and proliferation of superficial dermal capillaries following inflammatory acne lesions. It presents clinically as well-demarcated erythematous macules or patches, primarily located on previously inflamed sites. Although PAE can spontaneously resolve within 2 to 6 months, in many individuals-particularly those with darker Fitzpatrick skin types-it may persist significantly longer, often overlapping with post-inflammatory hyperpigmentation (PIH). Epidemiological data suggest that the incidence of PAE and PIH in darker-skinned populations ranges from 45.5% to as high as 87.2%, highlighting the need for effective interventions. Given that acne and its sequelae predominantly involve facial skin, the psychosocial burden is substantial. Patients often experience reduced self-esteem, social withdrawal, and even symptoms of anxiety and depression, underscoring the importance of timely and effective treatment strategies.

Among current therapeutic approaches, low-energy, large-spot 1064 nm Q-switched Nd:YAG laser has garnered attention due to its favorable safety profile and ability to penetrate deeper dermal layers. Operating in the near-infrared spectrum, the 1064 nm wavelength is selectively absorbed by hemoglobin in dilated capillaries, promoting vasoconstriction and diminishing visible erythema. At low energy densities, this laser minimizes thermal injury to surrounding tissues while simultaneously stimulating neocollagenesis, thereby contributing to both vascular remodeling and dermal regeneration. This dual mechanism supports its utility in managing PAE with minimal downtime.

In contrast, Delicate Pulsed Light (DPL), an advanced form of filtered intense pulsed light (IPL), offers enhanced precision through narrower wavelength bands, typically within the 500-650 nm range. This allows for more selective targeting of hemoglobin and melanin, improving therapeutic outcomes while reducing the risk of non-specific tissue damage. In the context of PAE, DPL effectively targets superficial vascular lesions, mitigates inflammatory processes, and promotes skin healing through controlled photothermal effects and collagen stimulation. Compared to conventional IPL, DPL provides improved treatment accuracy, reduced adverse effects, and better adaptability across a range of skin phototypes.

Given the growing demand for non-invasive, effective, and safe interventions for PAE, comparative studies on commonly used energy-based devices are warranted. Therefore, in this study, we conducted a prospective, split-face, randomized controlled trial to compare the clinical efficacy and safety of low-energy 1064 nm Nd:YAG laser and DPL in the treatment of acne and PAE. This design allows for intra-individual comparison, thereby minimizing confounding variables and enhancing the validity of outcome assessments. Our primary objective was to determine whether there are significant differences in the therapeutic outcomes between these two modalities, with a particular focus on erythema resolution, patient satisfaction, and adverse event profiles.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years, regardless of gender;
* Clinically and dermatoscopically diagnosed with acne and post-acne erythema (PAE) with bilaterally symmetrical facial lesions;
* Patients with normal cognitive function and stable mental status;
* Patients with good communication abilities;
* Voluntary participation in the study with signed informed consent.

Exclusion Criteria:

* Patients meeting any of the following conditions will be excluded from the study:
* History of photosensitivity;
* Presence of severe immunological disorders;
* Keloid or hypertrophic scarring tendency;
* Pregnant or breastfeeding individuals;
* Alcohol abuse;
* Presence of other facial skin diseases;
* Mental illness or psychiatric disorders that impair compliance;
* Currently pregnant or lactating;
* Presence of severe internal medical conditions;
* Poor treatment compliance or inability to cooperate due to psychiatric conditions.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2025-01-17 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
PAE lesion count | 0, 4, 8, 12 weeks
  The post-acne erythema (PAE) lesion count is an important objective indicator for assessing the severity of PAE. It involves recording the number of erythematous lesions on the face to evaluate changes before and after treatment. A higher lesion count indicates more severe erythema and poorer skin recovery. The assessment is typically conducted independently by two trained dermatologists under standardized lighting conditions, with high-resolution imaging systems used when necessary to enhance accuracy and consistency. Care is taken to distinguish PAE from other cutaneous manifestations such as active acne, post-inflammatory hyperpigmentation, and scarring. As a quantitative measure of erythema severity and improvement, the lesion count is widely applied in clinical studies involving light-based and laser therapies.

SECONDARY OUTCOMES:
CEA score | 0, 4, 8, 12 weeks
  The CEA score can be used to estimate the overall severity of the patient's condition. The score ranges from 0 to 4, with higher scores indicating more severe conditions.
erythema index | 0, 4, 8, 12 weeks
  Use non-invasive skin analyzer to measure the erythema index on the patient's facial skin at each follow-up visit.The larger the value, the more severe the erythema.
GFSS score | 0, 4, 8, 12 weeks
  The name of the scale is Global Flushing Severity Scale. The score ranges from 0 to 4, with higher scores indicating more severe conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Weihui zeng, Study Chair — Second Affiliated Hospital of Xi'an Jiaotong University
Locations (1):
- The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wu X, Wang X, Wu X, Cen Q, Xi W, Shang Y, Zhang Z, Lin X. Intense Pulsed Light Therapy Improves Acne-Induced Post-inflammatory Erythema and Hyperpigmentation: A Retrospective Study in Chinese Patients. Dermatol Ther (Heidelb). 2022 May;12(5):1147-1156. doi: 10.1007/s13555-022-00719-9. Epub 2022 Apr 12. PMID 35415801
- [Result] Urban K, Chu S, Giesey RL, Mehrmal S, Uppal P, Delost ME, Delost GR. Burden of skin disease and associated socioeconomic status in Asia: A cross-sectional analysis from the Global Burden of Disease Study 1990-2017. JAAD Int. 2020 Dec 10;2:40-50. doi: 10.1016/j.jdin.2020.10.006. eCollection 2021 Mar. PMID 34409353